CLINICAL TRIAL: NCT02168088
Title: Molecular Autopsy for Sudden Cardiovascular Death
Brief Title: Molecular Autopsy Study
Status: Recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, PI, Director STSI, Scripps Translational Science Institute
Other Study IDs: 14-6386
Record Dates: First submitted 2014-06-10; First posted 2014-06-20 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Sudden Unexplained Death
Keywords: Sudden unexplained death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and/or tissue will be collected on the deceased individual. Saliva samples will be collected on family members who have consented to participate.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Index case: Subjects who have died of sudden unexplained death
- Biologically related family member: Biologically related family member of the deceased individual

SUMMARY:
This study seeks to incorporate genetic testing into the postmortem examination of cases of sudden unexplained death.

DETAILED DESCRIPTION:
This study seeks to incorporate genetic testing into the postmortem examination of cases of sudden unexplained death, initially in San Diego County with plans to expand nationally and internationally as funding allows. Genetic testing of the index subjects and their parents (or other biological family members if parents are not available) will be assessed for potential heritable causes of sudden death. By combining the wide catchment base of the San Diego Medical Examiner's Office, sequencing expertise of SD-based collaborators, computing power of the San Diego Supercomputer Center and in-house and external genomic analytics, the Scripps Translational Science Institute aims to provide a more complete characterization and understanding of the genetic causes of sudden death. Ultimately, findings from this study will be utilized to identify previously unrecognized mechanism of sudden death allowing for the development of preventative screening programs and potentially life-saving interventions.

ELIGIBILITY:
Inclusion Criteria:

* Index case age between birth - 45 years
* Clinical presentation of sudden / unexplained death (believed to be cardiac in nature OR secondary to a massive unprovoked pulmonary embolism with no prior diagnosis of prothrombotic disease)

Exclusion Criteria:

* Premature death secondary to murder, suicide or external causal event
* Premature death thought secondary to known chronic comorbid medical condition
* Premature death thought secondary to end-organ failure (kidney, liver, lung) other than heart
* Previously diagnosed with hypertrophic cardiomyopathy (HCM)
* Prior myocardial infarction (regardless of stenting or bypass)
* Prior cerebrovascular accident (stroke or TIA)
* History of open heart surgery (for any reason)
* History of severe, untreated hypertensive heart disease
* History of illicit drug use
* History of heavy alcohol abuse
* History of severe pulmonary disease
* History of morbid obesity

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is limited to cases of sudden unexplained death in San Diego County and their living, biologically-related family members.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2025-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Heritable causes of sudden death | 3 years
  The primary endpoint for this study is the discovery of genomic information that may help identify a potential cause of death in the index case. This information may inform living, biologically related family members of their potential risk and need for further genomic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States